CLINICAL TRIAL: NCT02343328
Title: Placebo Controlled Study of Fecal Microbiota Transplant (FMT) for a First or Second Episode of C. Difficile Infection in Adults Using a Frozen Encapsulated Inoculum
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Not enough interest
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Elizabeth L. Hohmann, MD, Associate Professor of Medicine, Massachusetts General Hospital
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2014P002706
Record Dates: First submitted 2015-01-15; First posted 2015-01-22 (Estimated); Last update posted 2017-09-13 (Actual); Status verified 2017-09

CONDITIONS: Clostridium Difficile
MeSH Terms: interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Fecal Microbiota Transplant Capsules (Active Comparator): Fecal microbiota transplant capsules
  Interventions: Biological: Fecal Microbiota Transplant; Biological: Placebo
- Placebo Capsules (Placebo Comparator): Placebo capsules made from a mixture of natural cocoa powder and gelatin
  Interventions: Biological: Fecal Microbiota Transplant; Biological: Placebo

INTERVENTIONS:
Biological: Fecal Microbiota Transplant
Biological: Placebo

SUMMARY:
The investigators wish to compare Fecal Microbiota Transplant (FMT) capsules to placebo capsules in subjects with TWO episodes of C. difficile. The investigators have numerous subjects and physicians requesting FMT at the time of a second relapse, in order to prevent further hospitalizations, obtain a faster and more durable cure, avoid costly medications like fidaxomicin and oral vancomycin, and "fix" the underlying dysbiosis. In some instances, subjects feel like they are being asked to "get sick again" before they can pursue the most effective option. The investigators propose to study these subjects with a rigorous placebo controlled design, which will contribute significantly to our understanding of the utility of FMT, timing, and the real relapse rates in a tertiary referral center. Subjects who relapse with placebo will by definition have a third episode, meet consensus criteria for FMT, and will be offered "standard" FMT by capsule at that time. Additionally, this study will allow us to further capture safety data, in comparison to placebo capsules and further enhance our understanding of the microbiology of dysbiosis, earlier on in the illness course. Lastly, the investigators may decide to perform a cost analysis.

ELIGIBILITY:
Inclusion Criteria:

* Patients with two episodes of Clostridium dificile infection defined as having resolved symptoms after an initial microbiologically confirmed diagnosis of C. difficile, who have completed a course of antibiotics, and have a second positive test (toxin or PCR) obtained for a relapse of diarrhea symptoms by treating providers. Subjects with a positive "test of cure" stool sample (NOT advised by SHEA guidelines) in the absence of relapsed symptoms of CDI, or those who never improved their symptoms on the initial course of antibiotics will not be eligible. (Subjects who do not have a response to antibiotics may have other or additional diagnoses which are not likely to be helped by FMT.)
* Willingness to accept risk of unrelated donor stool.
* Age 18 or above. We do not believe there is a reason to have an upper age limit as long as patients can consent and can swallow large capsules. The elderly are disproportionately affected by CDI in terms of incidence, severity and affect on quality of life given limited mobility.
* Able to consent for self.
* Subjects are not expected to receive additional antibiotics for other indications in the next 8 weeks.
* Patients on a standard chemotherapeutic regimen for solid tumors, where significant duration of neutropenia is NOT expected in the 2 weeks following FMT may be enrolled with the agreement of their oncologist.
* Pt must be willing to have baseline Hepatitis B and C screening, and HIV screening (as required by the FDA for past studies). Those known to be seropositive for any of these illnesses need not be retested. These illnesses do not exclude subjects a priori, we simply wish to document initial sero-status.
* Subjects who have completed a second course of antibiotics may be enrolled up to 7 days after completing their second course of antibiotics for C. difficile

Exclusion Criteria:

* Delayed gastric emptying syndrome
* Known chronic aspiration
* Swallowing dysfunction or oral-motor dyscoordination, or inability or unwillingness to swallow multiple large capsules
* Pregnant women; we have previously and will continue to include postpartum and breastfeeding women. Women of child bearing potential have a urine or serum human chorionic gonadotropin test at enrollment.
* Patients with an acute illness unrelated to CDI or an acute exacerbation of underlying co-morbid condition
* Neutropenia (ANC <500) currently or expected within 2 weeks of FMT. (must have count within 7 d in relevant subjects, i.e. those with recent chemotherapy)
* Subjects on high dose steroids (>40 mg daily)
* Subjects on multiple/combination immunosuppressive regimens including high dose corticosteroids, calcineurin inhibitors, lymphocyte depleting biologic agents, anti-tumor necrosis factor agents. Subjects on a stable dose of a SINGLE immunosuppressive agent like steroids, rituximab, infliximab, other anti-TNF agents, with approval of the treating physician may be enrolled. These subjects may be at greatest risk of complications and hospitalization if another relapse of CDI occurs and may benefit.
* Patients with decompensated cirrhosis, advanced HIV/AIDS, recent bone marrow transplant, other cause of severe immunodeficiency.
* Patients with a history of significant allergy to foods not excluded from the donor diet (excluded foods are tree nuts, peanuts, shellfish, eggs)
* Ongoing systemic antibiotics for other infections (these people are better maintained on suppressive vancomycin and transplanted later). Subjects may have recently completed a course of antibiotics for another indication.
* Advanced HIV/AIDS with cluster of differentiation 4 cells (CD4) count less than 50.
* Allergy to chocolate/cocoa or gelatin, or unwillingness to ingest gelatin (in placebo capsules).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2015-01; Primary Completion 2016-07-29 (Actual); Study Completion 2016-07-29 (Actual)

PRIMARY OUTCOMES:
Resolution of diarrhea/Clostridium dificile infection symptoms and/or no relapse of C.difficile at 8 weeks | 8 weeks
  The primary objective of this study is to evaluate the safety and efficacy of FMT, and the relapse rate compared to placebo at 8 weeks, with cure defined by the absence of diarrhea/CDI symptoms at 8 weeks. We are defining the absence of relapsed CDI at 8 weeks symptoms as a cure.

SECONDARY OUTCOMES:
Self-reported weight | Over 6 months
Subjective well-being/improvement per standardized health rating scales (general health and GI health; as described above and on CRF). | Over 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Hohmann, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Background] Youngster I, Russell GH, Pindar C, Ziv-Baran T, Sauk J, Hohmann EL. Oral, capsulized, frozen fecal microbiota transplantation for relapsing Clostridium difficile infection. JAMA. 2014 Nov 5;312(17):1772-8. doi: 10.1001/jama.2014.13875. PMID 25322359